CLINICAL TRIAL: NCT06966011
Title: Pain Management After Total Knee Arthroplasty: Incidence and Outcomes of Rebound Pain
Brief Title: Rebound Pain After Peripheral Nerve Blocks in Total Knee Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 2.02.2025-35892
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty; Postoperative Pain; Rebound Pain; Peripheral Nerve Block; Pain Management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to determine the incidence and clinical impact of rebound pain after peripheral nerve blocks in patients undergoing total knee arthroplasty. Rebound pain is defined as a sudden, severe pain (NRS ≥7) emerging after block resolution. Primary outcome is the incidence of rebound pain; secondary outcomes include pain severity, rescue analgesia use, nausea, vomiting, sleep quality, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* ASA physical status I to III
* Scheduled for elective unilateral total knee arthroplasty under spinal anesthesia
* Peripheral nerve block (PNB) planned as part of multimodal analgesia
* Ability to understand and provide written informed consent
* Willingness and ability to complete the postoperative pain diary

Exclusion Criteria:

* Known allergy or hypersensitivity to local anesthetics
* Contraindication to regional anesthesia
* ASA physical status IV or higher
* Neurological or psychiatric disorders interfering with study participation or pain reporting
* Use of anticoagulants or presence of coagulopathy
* Use of medications that may alter pain perception or rebound pain response
* Local infection at the block site
* Emergency surgeries
* Inability or unwillingness to complete the postoperative pain diary or follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 70 years who are scheduled for elective unilateral total knee arthroplasty under spinal anesthesia at a tertiary care hospital. All participants will receive peripheral nerve blocks as part of a standardized multimodal analgesia protocol. Patients must be physically and cognitively able to provide consent and complete a postoperative pain diary. Those with contraindications to regional anesthesia, allergies to local anesthetics, or significant comorbidities (ASA IV and above) will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Rebound Pain After Peripheral Nerve Block | Within 48 hours after surgery
  Rebound pain is defined as a sudden, severe increase in pain occurring after the resolution of peripheral nerve block, typically within 12-24 hours postoperatively. Pain intensity will be assessed using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain). A score of NRS ≥7 will be considered as severe pain. Patients will record pain scores in a pain diary, and incidence will be calculated as the proportion of patients meeting the rebound pain criteria.

SECONDARY OUTCOMES:
Sleep Quality | From 1 day before surgery to postoperative day 7
  Sleep quality will be assessed using a 6-item sleep questionnaire (scored 1-6, where 1 = best and 6 = worst sleep quality), covering the night before surgery and the first 7 nights postoperatively.
Patient Satisfaction with Pain Management | Postoperative day 7 (via telephone follow-up)
  Patients will rate their satisfaction with postoperative pain control on a 5-point Likert scale (1 = not at all satisfied, 5 = completely satisfied).
Total Rescue Analgesic Consumption | Within 48 hours after surgery
  The total dose of rescue opioid analgesics administered within the first 48 hours postoperatively will be recorded in milligrams.
Time to First Rescue Analgesia | Within 48 hours after surgery
  Time elapsed from the end of surgery to the first administration of rescue analgesia will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data due to institutional policies and patient confidentiality considerations.